CLINICAL TRIAL: NCT02345811
Title: A Bilateral Dispensing Clinical Trial of Sapphire Lens Against Senofilcon A Lens Over 2 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-01
Record Dates: First submitted 2015-01-14; First posted 2015-01-26 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-07

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sapphire (Experimental): Participants were randomized to wear the Sapphire lens pair for two weeks during the cross over study.
  Interventions: Device: Sapphire
- senofilcon A (Active Comparator): Participants were randomized to wear the senofilcon A lens pair for two weeks during the cross over study.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: Sapphire — silicone-hydrogel contact lens
  Arms: Sapphire
Device: senofilcon A — contact lens
  Arms: senofilcon A

SUMMARY:
To evaluate the clinical performance of an investigational silicone-hydrogel lens when worn on a daily wear modality over two weeks of lens wear.

DETAILED DESCRIPTION:
This was a randomized, bilateral, 2 week cross over, double-masked, dispensing study comparing Sapphire test lens against the senofilcon A control lens. This study results were not used to support design validation of the test lens.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age for Canada and 18 years of age for the USA and has full legal capacity to volunteer
* Has read and signed an information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is an adapted soft contact lens wearer
* Requires spectacle lens powers between -0.50 to -6.00 diopters sphere (0.25D steps) or +1.00 to +8.00 diopters sphere (1.00D steps)
* Has no more than 0.75 diopters of refractive astigmatism
* Willing to wear contact lens in both eyes
* Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/25 in each eye
* To be eligible for lens dispensing, the subject must have VA of logMAR equivalent of 20/30 or better in each eye with the study lenses and the investigator must judge the fit as acceptable

Exclusion Criteria:

* Is participating in any concurrent clinical or research study
* Has any known active* ocular disease and/or infection
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit)
* Is aphakic
* Has undergone refractive error surgery

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lin, OD PhD, Principal Investigator — University of California, Berkeley; Lyndon Jones, PhD FCO, Principal Investigator — University of Waterloo CCLR
Locations (2):
- Clinical Research Center, University of California, Berkeley, Berkeley, California, United States
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Sapphire Lens Then Senofilcon A: Participants were randomized to wear the Sapphire lens pair for two weeks then cross over to Senofilcon A pair for two weeks.
  Sapphire Lens: silicone-hydrogel contact lens senofilcon A: contact lens
- Senofilcon A Then Sapphire Lens: Participants were randomized to wear the senofilcon A lens pair for two weeks then cross over to Sapphire lens pair for two weeks.
  senofilcon A: contact lens Sapphire lens: silicone-hydrogel contact lens
Period: First Intervention
Arm/Group | Sapphire Lens Then Senofilcon A | Senofilcon A Then Sapphire Lens
Started | 17 | 17
Completed | 16 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Sapphire Lens Then Senofilcon A | Senofilcon A Then Sapphire Lens
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear either the test lens or the control lens for 2 weeks and then cross-over to the other lens.
  Test Lens: Sapphire (contact lens) Control Lens : Senofilcon A (contact lens)
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 15
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Vision Quality
Description: Subjective rating for vision quality. Collected at dispense after settling of each study pair. (0-100 scale; 0=extremely poor vision, 100=excellent vision)
Time Frame: Baseline (10 minutes post lens settling at dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 93 (9) | 94 (7)

2. Primary Outcome: Vision Quality
Description: as for outcome 1
Time Frame: 2 weeks - During the Day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sapphire: Participants were randomized to wear the Sapphire lens pair for two weeks during the cross over study.
  Sapphire Lens: silicone-hydrogel contact lens
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 88 (12) | 91 (11)

3. Primary Outcome: Vision Quality
Description: as for outcome 1
Time Frame: 2 weeks - End of Day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 86 (14) | 87 (14)

4. Primary Outcome: Subjective Rating for Comfort.
Description: Subjective rating for comfort. Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever
Time Frame: Baseline - 10 minutes post lens settling
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 91 (12) | 92 (11)

5. Primary Outcome: Subjective Rating for Comfort.
Description: Subjective rating for comfort. Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever
Time Frame: 2-weeks - During the Day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 76 (20) | 87 (13)

6. Primary Outcome: Subjective Rating for Comfort.
Description: Subjective rating for comfort. Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever
Time Frame: 2-weeks - End of Day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 66 (26) | 81 (17)

7. Primary Outcome: Lens Surface Wettability
Description: Lens surface wettability assessed. Scale 0-4, 0.25 steps, 0=nonwetting, 4=excellent)
Time Frame: Baseline (10 minutes post lens settling)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
Number analyzed (Eyes) | 64 | 64
units on a scale | 3.2 (0.6) | 3.2 (0.7)

8. Primary Outcome: Lens Surface Wettability
Description: Lens surface wettability assessed. Scale 0-4, 0.25 steps, 0=nonwetting, 4=excellent)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
Number analyzed (Eyes) | 64 | 64
units on a scale | 3.0 (0.8) | 3.2 (0.6)

9. Primary Outcome: Surface Deposits
Description: Surface deposits is assessed. (Scale 0-4,0.25 steps) (0=no deposits; 1 = <5 deposits; 2 = >5 deposits or film 25-50% of surface; 3 = deposits 0.1 - 0.5mm or film 50-75% of surface; 4 = deposits >0.5mm or film > 75% of surface)
Time Frame: Baseline (10 minutes post lens settling)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 0.05 (0.18) | 0.16 (0.40)

10. Primary Outcome: Surface Deposits
Description: as for outcome 9
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 0.45 (0.51) | 0.40 (0.51)

11. Primary Outcome: Lens Handling (Ease of Insertion)
Description: Lens handling - ease of insertion of the lenses. Scale 0-100, 0=could not place lens on eye, 100=always easy to place lens on eye.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 93 (10) | 95 (8)

12. Primary Outcome: Lens Handling (Ease of Removal)
Description: Lens handling - ease of removal of the lenses. Scale 0-100, 0=could not remove lens from eye, 100=always easy to remove lens from eye.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire | Senofilcon A
Number analyzed (Participants) | 32 | 32
units on a scale | 90 (14) | 95 (7)

13. Primary Outcome: Subjective Preference for Comfort.
Description: Subjective rating for comfort. Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever
Time Frame: Baseline - 10 minutes post lens settling
Measure: Number; unit: percentage of participants
Groups:
- Overall Study: Participants were randomized to wear the Sapphire lens pair for two weeks and senofilcon A lens pair for two weeks during the cross over study.
  Sapphire: silicone-hydrogel contact lens senofilcon A: silicone-hydrogel contact lens
Arm/Group | Overall Study
Number analyzed (Participants) | 32
percentage of participants
  Sapphire | 22
  senofilcon A | 53
  No preference | 25

14. Primary Outcome: Subjective Preference for Comfort.
Description: Subjective rating for comfort. Scale 0-100, 0=cannot be worn, causes pain, 100=cannot be felt ever
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 32
percentage of participants
  Sapphire | 23
  senofilcon A | 68
  No preference | 9

ADVERSE EVENTS:
Time Frame: From dispense up to 2 weeks for each study lenses, a total of 4 weeks
Arm/Group | Sapphire | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 2/32 | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sapphire (N=32) | Senofilcon A (N=32)
Sore Throat and Fever (Infections and infestations) | 2 (2) | 0 (0)
Corneal Staining (Eye disorders) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No